CLINICAL TRIAL: NCT05610995
Title: Feasibility Study of Early Return-home After Colorectal Surgery Using a SENSIUM® Vital Parameter Monitoring Device
Acronym: Colo-SENSIUM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment faisibility
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 38RC21.0379
Record Dates: First submitted 2022-09-20; First posted 2022-11-09 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Premature Exit After Colorectal Surgery

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, randomized, two-arm, parallel, open-label, interventional controlled trial with masked outcome assessment (PROBE design)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SENSIUM Group (Experimental): Patients in the experimental group will be discharged with the device after an assessment on Day 1.
  Interventions: Device: SENSIUM Patch
- ERAS standard Group (No Intervention): Patients in the control group will receive the usual ERAS (conventional hospitalization for clinicobiological monitoring).

INTERVENTIONS:
Device: SENSIUM Patch — The SENSIUM device is a tool to monitor vital signs by applying a connected skin patch whose objective is to detect complications early. The health data is transmitted to the practitioner and in case of disturbance of the parameters, an alert is sent. The patient can be called for consultation or hospitalization if necessary. This device has been tested under real clinical conditions in surgical units. The continuous monitoring of vital signs resulted in earlier detection of sepsis, earlier administration of antibiotics, shorter average length of stay and lower 30-day readmission rates.
  Arms: SENSIUM Group

SUMMARY:
The principal aim of this study is to evaluate the impact on length of stay of a return-to-home monitoring device versus enhanced rehabilitation after bowel resection surgery with anastomosis.

The device SENSIUM is a tool to monitor vital signs (respiratory rate, heart rate and temperature) by applying a connected skin patch in order to detect complications early.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. ASA score 1-3
3. Colonic or rectal resection with anastomosis
4. Minimally invasive surgery
5. Patient living close to the hospital (<1 hour drive)
6. Patient accompanied for 48 hours
7. Body Mass Index < 40
8. Patient information and signature of consent
9. Patient affiliated to a social insurance plan
10. A pregnancy test must be performed before inclusion in women of childbearing age.

Non-inclusion Criteria:

1. Socially isolated patient and/or no 3G cell signal
2. Severe comorbidities defined as any of these characteristics:

   1. Severe malnutrition (albumin <30g/l)
   2. Severe anemia < 80 g/dl
   3. Insulin-dependent diabetes type 1

   e. Patient under anticoagulation f. Severe renal insufficiency
3. History of psychiatric illness with medication requirements
4. Persons referred to in articles L1121-5 to L1121-8 of the CSP (corresponds to all protected persons: pregnant women, parturients, nursing mothers, persons deprived of liberty by judicial or administrative decision, persons under legal protection)
5. Patient not wishing to enter the study
6. Patient in a period of exclusion from another study or ongoing participation in an interventional study

Exclusion Criteria:

1. Stoma preparation
2. Per operative conversion to laparotomy
3. CHUNG score > 8

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-07-22 (Actual); Primary Completion 2024-10-08 (Actual); Study Completion 2024-10-08 (Actual)

PRIMARY OUTCOMES:
Evaluating the impact on length of stay of a return-to-home monitoring device versus enhanced rehabilitation after bowel resection surgery with anastomosis | at Day 30
  Overall length of stay of the patient (index stay, and possible re-hospitalizations)

SECONDARY OUTCOMES:
Assess transit recovery | at Day 1
  Time of resumption of transit formalized by the resumption of gas, the time being calculated between the closure of the skin and the first gas in hours
Assess pain | at Day 0, Day 1, Day 2, Day 3, Day 4, Day 5 and Day 30
  Pain, by visual analog scale (0-10)
Assess opioid use | at Day 5
  5-day opioid consumption rate
Evaluate the complication rate | at Day 30 according to the postoperative management performed
  Presence of a complication according to the Clavien Dindo classification
Evaluate the rate of re-hospitalization performed | To the post-surgical hospital discharge at Day 30
  Presence of a rehospitalization between the post-surgical hospital discharge and Day 30
Assess the rate of unscheduled visits | at Day 30
  Presence of an unscheduled consultation at Day 30 post-surgery
Assess the patient's quality of life and overall satisfaction | at Day 30
  EuroQol 5D 3L standardized scale score (overall satisfaction) at pre-inclusion, Day 1, Day 5 and Day 30 post-surgery visit
Evaluate the cost of care | To Day 1 at the end of study
  Cost analysis (hospitalizations, consultations, re-interventions, time off work, transportation and SENSIUM system costs)
Evaluate the evolution of vital parameters | To Day 1 at the end of study
  Trend analysis of vital parameters

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Chu Amiens, Amiens
  - CHU Angers, Angers
  - Clinique TIVOLI, Bordeaux
  - Chru Brest, Brest
  - CHU Grenoble Alpes, Grenoble
  - Institut Paoli Calmettes, Marseille
  - Chu Nantes, Nantes